CLINICAL TRIAL: NCT00561431
Title: A Randomized Prospective Study Comparing High Dose Continuous Venovenous Hemodiafiltration (CVVHDF) to Standard Dose CVVHDF in Critically Ill Patients With Acute Renal Failure at the University of Alabama at Birmingham
Brief Title: High Dose CVVHDF Compared to Standard Dose CVVHDF
Acronym: CVVHDF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ashita Tolwani, Principal Investigatorl, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X030108004
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Acute Renal Failure
Keywords: CVVHDF Dose Study
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Standard dose Continuous Venovenous Hemodiafiltration (CVVHDF) at an effluent rate of 20 ml/kg/hr
  Interventions: Device: Standard dose of dialysis
- 2 (Experimental): High dose Continuous Venovenous Hemodiafiltration (CVVHDF) at an effluent rate of 35 ml/kg/hr
  Interventions: Device: High dose of dialysis

INTERVENTIONS:
Device: Standard dose of dialysis — Continuous Venovenous Hemodiafiltration (CVVHDF) effluent dose of 20 ml/kg/hr
  Arms: 1
Device: High dose of dialysis — Continuous Venovenous Hemodiafiltration (CVVHDF) effluent rate 35 ml/kg/hr
  Arms: 2

SUMMARY:
In the last three decades, the mortality associated with acute renal failure (ARF) in the ICU has remained unchanged at greater than 50%, despite improvements in dialysis technology.

The primary objective is to determine whether Continuous Veno-Venous Hemodiafiltration (CVVHDF) using an ultrafiltration rate of 35 ml/hr/kg (high dose) leads to a greater reduction in all-cause ICU mortality compared to standard CVVHDF using an ultrafiltration rate of 20 ml/hr/kg.

DETAILED DESCRIPTION:
Although the worldwide standard for renal replacement therapy is intermittent hemodialysis(IHD), continuous renal replacement therapy (CRRT) has emerged as an alternative form of renal replacement therapy in the critical care setting due to its advantages of slow continuous fluid removal, steady acid-base correction, and hemodynamic stability.

There are no standard protocols for initiating or administering CRRT, and practice patterns vary widely among institutions, with less than 25% of patients with ARF in the ICU receiving this therapy in the United States.

Various CRRT modalities are available that use diffusion, convection, or a combination of both to obtain adequate solute clearance. However, there is no consensus as to the optimal dialysis modality, adequate dialysis dose, or optimal clearance modality (convection vs. diffusion). Clinical trials are needed to determine the optimal method of administering CRRT, with respect to modality, dose of dialysis, and time of initiation of therapy.

Although some studies suggest that a higher dose of dialysis improves survival, there have been no prospective randomized studies comparing the effectiveness of diffusion and convection, combined together, for solute clearance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > or equal to 19 yrs of age
* ARF defined by at least one of the following:

  * Volume overload from inadequate urine output despite diuretic agents.
  * Oliguria (urine output < 200 ml/12hrs) despite fluid resuscitation and diuretic administration.
  * Anuria (urine output < 50 ml/12 hrs).
  * Acute azotemia (BUN > or equal to 80 mg/dl).
  * Acute hyperkalemia not responsive to medication (K+ > or equal to 6.5mmol/L)
  * An increase in serum creatinine of > 2.5 mg/dl from normal values or a sustained rise in serum creatinine of > or equal to 1 mg/dl over baseline.

Exclusion Criteria

* Patients with end stage renal disease
* Patients who have had more than one previous dialysis session for acute or chronic renal failure during the current hospitalization
* Patient weight greater than 125 kg
* Patient weight less than 50 kg
* Pregnancy
* Prisoner
* Non-candidacy for continuous renal replacement therapy (CRRT)
* Patient/surrogate refusal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashita J. Tolwani, MD, Principal Investigator — The University of Alabama at Birmingham, Division of Nephrology
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF): Standard dose Continuous Venovenous Hemodiafiltration (CVVHDF) at an effluent rate of 20 ml/kg/hr
- High Dose Continuous Venovenous Hemodiafiltration (CVVHDF): High dose Continuous Venovenous Hemodiafiltration (CVVHDF) at an effluent rate of 35 ml/kg/hr
Period: Overall Study
Arm/Group | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF)
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 64 | 121
  >=65 years | 43 | 36 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15) | 58 (16) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 57 | 59 | 116
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive at 30 Days After Enrollment Compared Between High Dose Versus Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF)
Description: The primary objective is to determine whether Continuous Venovenous Hemodiafiltration (CVVHDF) using an effluent rate of 35 ml/hr/kg (high dose) leads to an increased participant survival time as compared to CVVHDF using the standard effluent rate of 25 ml/hr/kg as measured by days on continuous renal replacement therapy (CRRT) at enrollment up to 30 days.
Time Frame: Up to 30 days
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF)
Number analyzed (Participants) | 100 | 100
participants | 56 | 49

2. Secondary Outcome: Recovery of Renal Function, Defined as Not Requiring Dialysis After Discontinuation of CRRT
Description: The number of participants who recover renal function at 30 days after enrollment in each arm.
Time Frame: Up to 30 days
Population: intention to treat
Measure: Number; unit: Participants
Arm/Group | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF)
Number analyzed (Participants) | 100 | 100
Participants | 37 | 28

ADVERSE EVENTS:
Time Frame: Time on continuous venovenous hemodiafiltration up to 30 days.
Description: The adverse events of death and non renal recovery were not related to the intervention or unexpected. The therapy did not affect this outcome.
Arm/Group | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF)
Serious Adverse Events (participants affected / at risk) | 63/100 | 72/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Dose Continuous Venovenous Hemodiafiltration (CVVHDF) (N=100) | High Dose Continuous Venovenous Hemodiafiltration (CVVHDF) (N=100)
death (General disorders) | 44 (44) | 51 (51)
Renal Failure (Renal and urinary disorders) | 63 (63) | 72 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No